CLINICAL TRIAL: NCT04462107
Title: Longitudinal Study Evaluating Postpartum Recovery After Scheduled Cesarean Delivery With the Obstetric Quality of Recovery Tool
Brief Title: Longitudinal Study Evaluating Recovery After Scheduled Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emily E. Sharpe, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 19-012077
Record Dates: First submitted 2020-04-07; First posted 2020-07-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surveys: All participants will complete questionnaires at several time points, ranging from baseline to 3 months post partum.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — All participants will complete surveys that range in time from baseline to 3 months post partum.

SUMMARY:
The purpose of this research is to describe how patients recover after scheduled C-section for the first 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older who receive neuraxial anesthesia for elective cesarean delivery

Exclusion Criteria:

* Less than 18 years of age
* Gestational age less than 32 weeks
* Women whose infants have died or are in the neonatal intensive care unit after delivery
* Inability to read or understand written English
* Failed neuraxial anesthesia requiring general anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women whom are pregnant and will have a scheduled C-section to deliver infant
Study Population: Parturients scheduled for cesarean delivery at Mayo Clinic Hospital Family Birth Center
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal evaluation of global health visual analog scale | Baseline, 24 h, 48 h, 1 week, 3 weeks, 6 weeks, 12 weeks postpartum
  Global health on a scale of 0-100 to indicate current health status with 0 being the worst imaginable health and 100 being the best health imaginable. Plan was to identify the plateau of improvement of GHVAS postpartum.

SECONDARY OUTCOMES:
To determine change in pain levels post C-section using the Visual Analog Scale (VAS) | Baseline, 24 hour, 48 hour, 1 week, 3 weeks, 6 weeks, 12 weeks, and 3 months
  Describes pain from no pain at all to the worst pain imaginable using a 100mm horizontal line
Compare opioid consumption post partum | 24 hours, 48 hours, 1 week, 3 weeks, 6 weeks, and 3months post partum
  Compare opioid consumption post partum
Compare non-maternal reasons for delayed hospital discharge | Hospital discharge, approximately 3 days
  Document non-maternal reasons for delayed hospital discharge such as NICU admission of neonate, neonatal IV antibiotics, delay in transportation, delay from pediatric team.
Compare frequency of activities of daily living | Baseline
  Activities of daily living are routine activities people do everyday without assistance including eating, bathing, getting dressed, toileting, cooking, cleaning, driving, shopping. Subject will report these activities as not done yet, done once, once/week, do most days, do every day
Compare frequency of activities of daily living | 6 weeks postpartum
  Activities of daily living are routine activities people do everyday without assistance including eating, bathing, getting dressed, toileting, cooking, cleaning, driving, shopping. Subject will report these activities as not done yet, done once, once/week, do most days, do every day
Compare Edinburgh Postnatal Depression Scale | 6 weeks postpartum
  Edinburgh Postnatal Depression Scale is a 10 item questionnaire to identify women who have postpartum depression
Compare a modified recovery after delivery questionnaire | 6 weeks postpartum
  9 questions that ask the mother about feeding baby, sleep, fatigue, bonding, parenting, and social functioning
Correlation between postpartum ObsQOR-10 and EQ-5D | 6 weeks postpartum
  EQ-5D describes current health for mobility, self-care, usual activities, pain, anxiety and on a scale of 0-100 to indicate current health status with 0 being the worst imaginable health and 100 being the best health imaginable. The ObsQOR-10 uses a scale of 0-10 with 0 being none and 10 being the worst imaginable, scoring pain, nausea, dizziness, shivering, comfort level, mobilization, holding baby, feeding baby, personal care, and feeling in control.
Correlation between postpartum ObsQOR-10 and EQ-5D | 12 weeks postpartum
  EQ-5D describes current health for mobility, self-care, usual activities, pain, anxiety and on a scale of 0-100 to indicate current health status with 0 being the worst imaginable health and 100 being the best health imaginable. The ObsQOR-10 uses a scale of 0-10 with 0 being none and 10 being the worst imaginable, scoring pain, nausea, dizziness, shivering, comfort level, mobilization, holding baby, feeding baby, personal care, and feeling in control.
Correlation between ObsQOR-10 scores at multiple time points | 24 hours, 48 hours, 1 week postpartum
  The ObsQOR-10 uses a scale of 0-10 with 0 being none and 10 being the worst imaginable, scoring pain, nausea, dizziness, shivering, comfort level, mobilization, holding baby, feeding baby, personal care, and feeling in control.
Correlation between postpartum ObsQOR-10 and EQ-5D | 3 weeks post partum
  EQ-5D describes current health for mobility, self-care, usual activities, pain, anxiety and on a scale of 0-100 to indicate current health status with 0 being the worst imaginable health and 100 being the best health imaginable. The ObsQOR-10 uses a scale of 0-10 with 0 being none and 10 being the worst imaginable, scoring pain, nausea, dizziness, shivering, comfort level, mobilization, holding baby, feeding baby, personal care, and feeling in control.

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Sharpe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Sharpe EE, Sviggum HP, Carvalho B, Guo N, Arendt KW, Stoltenberg AD, Tinaglia AG, Torbenson VE, Sultan P. Profiling Postpartum Recovery After Scheduled Cesarean Delivery With Neuraxial Anesthesia: A Longitudinal Cohort Study. Anesth Analg. 2025 Nov 1;141(5):1089-1096. doi: 10.1213/ANE.0000000000007476. Epub 2025 Apr 4. PMID 40184308
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials